CLINICAL TRIAL: NCT04227860
Title: The Effect of Combined Balance and Strength Exercise Program in Patients With Different Grades of Primary Knee Osteoarthritis Patients
Brief Title: Balance and Strength Exercise in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Yousra Hisham Abdel Fattah, Lecturer of Physical Medicine, Rheumatology and Rehabilitation, University of Alexandria
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0105852
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Post-exercise training assessment will be done by an investigator not involved in the study and unaware of the grading of KOA or of the pre-exercise assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: G I primary KOA (Active Comparator): Exercise and balance training
  Interventions: Other: Balance exercise program; Other: Strengthening exercise program
- Group 2: G II primary KOA (Active Comparator): Exercise and balance training
  Interventions: Other: Balance exercise program; Other: Strengthening exercise program
- Group 3: G III primary KOA (Active Comparator): Exercise and balance training
  Interventions: Other: Balance exercise program; Other: Strengthening exercise program
- Group 4: G IV primary KOA (Active Comparator): Exercise and balance training
  Interventions: Other: Balance exercise program; Other: Strengthening exercise program

INTERVENTIONS:
Other: Balance exercise program — Patients will be engaged in lower extremity kinesthesia and balance exercise program 3 time per week for 6 weeks.
  Divided into 2 stages, stage 1 and 2, each stage 3 weeks. Patients who fulfill at least stage 1 of the program will be included in the study.
Other: Strengthening exercise program — Patients will be engaged in strengthening exercise program 3 time per week for 6 weeks.
  Divided into 3 stages, stage 1, 2 and 3, each stage 2 weeks. Patients who fulfill at least stage 1 of the program will be included in the study.

SUMMARY:
The aim of this study is to assess the effect of balance exercise on dynamic balance and physical function in 80 patients with different grades of primary knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
The study will include 80 patients with primary knee osteoarthritis divided into 4 groups according to the Kellgren and Lawrence grading scale (KL):

Group 1: 20 patients with grade I KOA Group 2: 20 patients with grade II KOA Group 3: 20 patients with grade III KOA Group 4: 20 patients with grade IV KOA

* Patients will undergo pre-exercise and post- exercise assessment with:

  1. Western Ontario and McMaster University Osteoarthritis Index (WOMAC)
  2. Modified Stare Excursion Balance test
  3. Timed up and Go test
* Exercise program includes:

  1. Lower extremity kinesthesia and balance exercise program
  2. Strength exercise program

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthritis according to the EULAR recommendations 2010.
* Patients can complete at least stage 1 of balance and exercise program (minimum of 2 weeks)

Exclusion Criteria:

* Patients that cannot complete at least stage 1 of balance and exercise program
* Patients with medical conditions affecting postural balance including visual, inner ear and neurological problems.
* Patients with lower limb joint or bony problems other than primary knee osteoarthritis .
* Patients with secondary KOA.
* Patients who received intra- articular joint injection in 1 or both knees in the past 90 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | 2-6 weeks
  Using the Western Ontario and McMaster University Osteoarthritis Index (WOMAC), which contains pain sub-score and a overall total score. The higher the score the worst the pain.
Assessment of stiffness | 2-6 weeks
  Using the Western Ontario and McMaster University Osteoarthritis Index (WOMAC), which contains stiffness sub-score and a overall total score. The higher the score the worst the stiffness.
Assessment of physical function | 2-6 weeks
  Using the time up and go test, where the patient is seated and asked to get up walk a distance turn around and return to chair and sit again. It is measured using a timer, the longer the patient takes the worst the physical function of the patient.

SECONDARY OUTCOMES:
Dynamic Balance | 2-6 weeks
  Using the Modified star excursion balance test which measures the patients dynamic balance in several directions, giving the patient 3 attempts and measuring each time and taking a mean of the 3 measurements in each. An increase in the measurements means better dynamic balance and a smaller measurement means worse dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Yousra H Abdel Fattah, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No